CLINICAL TRIAL: NCT02091518
Title: Development and Evaluation of Magnetic Resonance Imaging Acquisition and Analysis Methods
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ceretype (Unknown); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-239
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: MRI; 13-239; volunteers; patients

ARMS (1):
- MRI (Experimental): Add-On Research Patients will include patients who are scheduled for a routine clinical MRI who meet the eligibility requirements for this protocol. Protocol participation will consist of an "add-on" research. MRI scan, which will be performed any point during of the routine clinical MRI scan.
  Volunteers will be subjects expressing interest in participation and who meet the eligibility requirements for this protocol. No contrast enhanced research MRIs including gadolinium-based or other contrast agents will be performed in volunteers.
  Interventions: Behavioral: MR Screening Questionnaire; Device: Magnetic Resonance Imaging Acquisition and Analysis

INTERVENTIONS:
Behavioral: MR Screening Questionnaire — All participants will complete the MR Screening Questionnaire before the MRI exam. During the MRI exam, all participants will be observed through the window from the operator console. Verbal communication will be kept with the participant throughout the exam via a speaker system.
Device: Magnetic Resonance Imaging Acquisition and Analysis — MRI Studies: The MRI scans will be performed on a 1.5T or 3T MRI scanner. Conventional MRI studies will be performed using the standard clinical sequences. The new research sequences will be performed.at any point during the clinical exam. Total imaging time for volunteers will be 30-45 minutes.

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic imaging method with constant progress and improvement in the way the MRI images are obtained. Many of these advances involve changes to MRI software and hardware. The goal of this study is to find out the possible benefits of new MRI techniques. This will allow us to use the new MRI methods in research and patient care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 or older

Exclusion Criteria:

* Anyone who would be normally excluded from undergoing an MRI examination as per Memorial Hospital for Cancer and Allied Diseases Screening Questionnaire for MRI
* Patients/volunteers with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field
* Female patients/ volunteers who are pregnant or nursing
* Patients/ volunteers who are unable to comply or complete the MRI exam due to claustrophobia or high levels of anxiety
* Patients/ volunteers from the vulnerable population, as defined by 45 CFR 46.
* Patients at higher risk due to age, frailty, or the emergent nature of their condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 461 (Estimated)
Dates: Start 2014-03; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
feasibility of new MRI applications | 5 years
  This protocol will provide pilot data to determine the feasibility of development and optimization of new MRI acquisition and analysis method.including sequence development, optimization, and workflow and analysis/visualization tools. An investigator will view the conventional images, as well as the additional research sequences. The radiologist will then complete data forms for each image and quantitative values, as listed in the evaluation form will be recorded. After all images have been read, the radiologist will review the clinical images together with the research images, and determine whether the research sequences had any effect on their diagnostic confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Akin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/